CLINICAL TRIAL: NCT03977129
Title: A Multicenter, Prospective, Randomized, Blind, Controlled Clinical Study to Compare the Efficacy of Quantitative Flow Ratio Guided and Coronary Angiography Guided Revascularization Strategy for Patients Undergoing Primary Valve Surgery With Comorbid Coronary Artery Disease
Brief Title: Quantitative Flow Ratio (QFR) Guided Coronary Artery Bypass Grafting for Patients Undergoing Primary Valve Surgery With Concomitant Coronary Artery Disease
Acronym: FAVOR IV-QVAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Med-X Research Institute, Shanghai Jiao Tong University (Unknown)
Responsible Party: Principal Investigator, Qiang Zhao,MD, Professor and Director, Department of Cardiovascular Surgery, Vice President, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018CR001
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Primary Valvular Heart Disease With Comorbid Coronary Artery Disease; Planned to Undergo Elective On-pump Valve Surgery Due to Primary Mitral and/or Aortic Valvular Heart Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QFR group (Experimental)
  Interventions: Device: QFR-guided strategy
- CAG group (Active Comparator)
  Interventions: Other: CAG-guided strategy

INTERVENTIONS:
Device: QFR-guided strategy — In this study, the QFR-guided strategy will be applied to in the QFR group in which calculation of the QFR values of all target coronary arteries with lesions with diameter stenosis of ≥ 50% (visual estimation) and with suitability to CABG revascularization will be carried out. If QFR ≤ 0.80, then simultaneous CABG revascularization of target blood vessels will be carried out. If QFR > 0.80, then no CABG revascularization of target blood vessels will be carried out.
  Arms: QFR group
Other: CAG-guided strategy — In this study, CAG-guided strategy will be used for the control group, i.e., in accordance with current guideline recommendations, all target coronary arteries with lesions with diameter stenosis of ≥ 50% (visual estimation) and suited for CABG revascularization will undergo CABG revascularization.
  Arms: CAG group

SUMMARY:
This is a multicenter, prospective, randomized, blinded, controlled clinical study in patients with planned primary valvular surgery and comorbid coronary artery lesions with diameter stenosis of ≥ 50%, to compare the effectiveness of an Quantitative Flow Ratio (QFR)-guided revascularization strategy and a coronary angiography (CAG)-guided revascularization strategy in preventing the incidence of composite outcome (MACE-5, including all-cause death, myocardial infarction, stroke, unplanned coronary revascularization, and new renal failure requiring dialysis) within 30 days after surgery. The study hypothesis is that the QFR-guided strategy can reduce the incidence of the MACE-5 within 30 days after surgery, as compared with the CAG-guided strategy.

DETAILED DESCRIPTION:
It is planned to enroll 792 subjects aged ≥18 years, with no gender restriction, who plan to undergo elective open-heart valvular surgery due to primary valvular heart disease, with comorbid coronary artery lesions defined as diameter stenosis of ≥ 50% (visual estimation) that are diagnosed by CAG before the surgery.

QFR group: Calculate the QFR values of all target coronary arteries (anterior descending branch, circumflex branch, main right coronary artery or its primary branches with ≥ 1.5 mm in diameter, such as diagonal branch, intermediate branch, obtuse marginal branch, posterior descending branch and posterior branch of left ventricle) with lesions with diameter stenosis of ≥ 50% (visual estimation) suited for CABG revascularization. If QFR ≤ 0.80, then simultaneous CABG revascularization of target blood vessels will be carried out. If QFR > 0.80, then no CABG revascularization of target blood vessels will be carried out.

CAG group (control group): All target coronary arteries (anterior descending branch, circumflex branch, main right coronary artery or its primary branches with ≥ 1.5 mm in diameter, such as diagonal branch, intermediate branch, obtuse marginal branch, posterior descending branch and posterior branch of left ventricle) with lesions with diameter stenosis of ≥ 50% (visual estimation) suited for CABG revascularization will undergo simultaneous CABG revascularization.

Intervention duration: The assessments will be performed after randomization and before the surgery to guide the surgery.

No planned interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the trial and provide the informed consent form;
* Male or female patients aged ≥ 18 years;
* Planned to undergo elective on-pump valve surgery due to primary mitral and/or aortic valvular heart disease (such as rheumatic, degenerative, infective, congenital valvular heart disease, etc.);
* At least one target coronary arteries (anterior descending branch, circumflex branch, main right coronary artery or its primary branches with ≥ 1.5 mm in diameter, such as diagonal branch, intermediate branch, obtuse marginal branch, posterior descending branch and posterior branch of left ventricle) with preoperative diameter stenosis of ≥ 50% by coronary angiography (visual estimation, subject to written coronary angiography report) and suited for CABG revascularization.

Exclusion Criteria:

* History of heart surgery;
* Planned second-stage PCI or CABG revascularization;
* Secondary valvular heart disease (ischemia, cardiomyopathy);
* Planned valve intervention surgery through the catheter;
* Subjects that were evaluated to have cardiogenic shock or other critical conditions that were not appropriate for the trial by study physician;
* QFR calculations cannot be carried out from preoperative coronary angiography data (such as poor projection position, inability to detect vascular boundaries, poor contrast agent filling, excessive overlap or severely distorted of vessel lesion sections, lesion involved in myocardial bridge, or lesion site within 3 mm from the ostium of the main coronary artery);
* The target coronary arteries were evaluated to be not suitable for CABG by study physician;
* Life expectancy < 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The 30-day incidence of composite outcome (MACE-5) including all-cause death, myocardial infarction, stroke, unplanned coronary revascularization, and new renal failure requiring dialysis | within 30 days after surgery

SECONDARY OUTCOMES:
The time from randomization to first occurrence of any of composite outcome (MACE-6) within 1 year | within 1 year after surgery
  The time from randomization to first occurrence of any of composite outcome (MACE-6) including all-cause death, myocardial infarction, stroke, unplanned coronary revascularization, hospitalization or urgent visits for unstable angina pectoris, and hospitalization or urgent visits for heart failure
The incidence of 1-year graft failure (stenosis ≥ 50% or occlusion occurred in grafts or distal anastomosis) | at 1 year after surgery
The time from randomization to first occurrence of any of composite outcome (MACE-6) within 3 year | within 3 years after surgery
  The time from randomization to first occurrence of any of composite outcome (MACE-6) including all-cause death, myocardial infarction, stroke, unplanned coronary revascularization, hospitalization or urgent visits for unstable angina pectoris, and hospitalization or urgent visits for heart failure
The incidence of 3-year graft failure (stenosis ≥ 50% or occlusion occurred in grafts or distal anastomosis) | at 3 years after surgery
Health-related quality of life | within 30 days, 1 year and 3 years after surgery
  the variables are the EQ-5D scores
Cost effectiveness | within 30 days, 1 year and 3 years after surgery
  the variables are the cost increased for each composite outcome reduction at 30 days after surgery and cost increased for each additional QALY at 1 year and 3 years after surgery

OTHER OUTCOMES:
The number of grafts per person | at Day 0
  counted as distal anastomosis
The total circulatory time during the surgery | at Day 0
  minutes
The total cross-clamp time during the surgery | at Day 0
  minutes
The total units of erythrocyte transfusion during and after the surgery till discharge | from Day 0 to discharge day
The number of days from surgery day to discharge day | from Day 0 to discharge day
Change from baseline in the Canadian Cardiac Society (CCS) anginal status score (0-4) | at 1 year after surgery
Change from baseline in the CCS anginal status score (0-4) | at 3 years after surgery
Change from baseline in the New York Heart Association (NYHA) score (1-4) | at 1 year after surgery
Change from baseline in the NYHA score (1-4) | at 3 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zhao, MD., Principal Investigator — Ruijin Hospital; Shengxian Tu, PhD., Principal Investigator — Med-X Research Institute, Shanghai Jiao Tong University; Yunpeng Zhu, MD., Study Director — Ruijin Hospital; Mario Gaudino, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (12):
- China (12):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second XiangYa Hospital of Central South University, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Zhu J, Zhu Y, Zhang W, Wang Z, Ye X, Zhou M, Li H, Qiu J, Xu H, Sun Y, Kang L, Tu S, Zhao Q. Preliminary outcomes of quantitative flow ratio-guided coronary bypass grafting in primary valve surgery: A propensity score weighted analysis. JTCVS Open. 2024 Jun 25;21:90-108. doi: 10.1016/j.xjon.2024.06.008. eCollection 2024 Oct. PMID 39534354